CLINICAL TRIAL: NCT03445936
Title: PRELOOP Trial: Synthetic Versus Biological Mesh for Prevention of Incisional Hernia After Loop-ileostomy Closure
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Elisa Mäkäräinen, MD, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 317/2017
Record Dates: First submitted 2018-02-07; First posted 2018-02-26 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Rectum Cancer
Keywords: loop-ileostomy reversal; hernia prevention
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized controlled multicenter trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Subject is blinded of the mesh used. Outcome at 10 month follow-up is assessed by surgeon who was not involved in the operation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parietene Macro (Active Comparator): Parietene Macro is a macroporous synthetic mesh used in retro muscular sublay position to prevent incisional hernia after loop-ileostomy closure.
  Interventions: Device: Parietene Macro
- Permacol (Active Comparator): Permacol is a acellular porcine dermal implant used in retro muscular sublay position to prevent incisional hernia after loop-ileostomy closure.
  Interventions: Device: Permacol

INTERVENTIONS:
Device: Parietene Macro — Parietene Macro is placed and sutured on retro muscular space on closed posterior rectus sheath to prevent incisional hernia.
  Arms: Parietene Macro
Device: Permacol — Permacol biologic implant is placed and sutured on retro muscular space on closed posterior rectus sheath to prevent incisional hernia.
  Arms: Permacol

SUMMARY:
This study compares a synthetic mesh and biological implant in prevention of incisional hernia after loop-ileostomy closure.

DETAILED DESCRIPTION:
Incisional hernia after loop-ileostomy closure may be an underestimated problem. Research on both biological and synthetic mesh in this context is scarce and no randomized controlled trials comparing meshes exist.

The aim of this study is to compare Parietene Macro and Permacol in prevention of incisional site hernia after temporary loop-ileostomy reversal after anterior resection and TME for rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Anterior resection and TME with temporary loop-ileostomy for rectal carcinoma
* 18 years or older
* Patient has a life expectancy of at least 12 months.
* Patient signs the Informed consent and agrees to attend all study visits

Exclusion Criteria:

* Patient with a comorbid illness or condition that would precluded the use of surgery (ASA 4-5).
* Patients with concurrent or previous malignant tumors within 5 years before study enrollment
* Patients with T4b tumors which imposed a multi-organ resection
* Patient undergone emergency procedures
* Primary rectal surgery along with major concomitant procedures (e.g. hepatectomies, other intestinal resections).
* Metastatic disease with life expectancy of less than 12 months
* Pregnancy or suspected pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-02-13 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Surgical site infection | 30 days
  The incidence of surgical site infections at 30 days follow up
Incisional hernia | 10 months
  Incidence of incisional hernia

SECONDARY OUTCOMES:
Complications classified by Clavien-Dindo classification | 30 days
  Clavien-Dindo I-V complications at 30 days follow-up
Re-operation rate | 5 years
  Demand for re-operations related to mesh or complications
Operative time | 30 days
  Time (min) needed for operation and application of mesh/implant
Length of stay | 30 days
  Length of stay at the hospital after the operation
Quality of life measured by RAND-36 survey | 5 years
  Quality of life after the operation measured by RAND 36
Incidence of hernia | 5 years
  Incidence of incisional hernia
Cost analysis | 5 years
  Analysis of costs to both individual and community

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Mäkäräinen-Uhlbäck, Principal Investigator — Oulu University Hospital
Locations (4):
- Finland (4):
  - Jyvaskyla Central Hospital, Jyväskylä
  - Oulu University Hospital, Oulu
  - Seinajoki Central Hospital, Seinäjoki
  - Tampere University Hospital, Tampere

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Makarainen EJ, Wiik HT, Kossi JAO, Pinta TM, Mantymaki LJ, Mattila AK, Nikki MJ, Jarvinen JE, Ohtonen PP, Rautio TT. Prevention of incisional hernia with retrorectus synthetic mesh versus biological mesh following loop ileostomy closure (Preloop trial). Br J Surg. 2024 Jan 3;111(1):znad362. doi: 10.1093/bjs/znad362. PMID 37944025